

College of Arts and Sciences Department of Psychology University of Cincinnati Cincinnati, OH, 45221

Official Title: Healthy Start to Feeding Pilot Trial

Brief Title: Healthy Start to Feeding Intervention

NCT Number: NCT03597061

Document Date: 7/9/2018

Date Uploaded: 6/24/21

Document: Statistical Analysis Plan



College of Arts and Sciences Department of Psychology University of Cincinnati Cincinnati, OH, 45221

## **Statistical Analysis Plan**

Primary Aim (Examine the impact of the HSF intervention on growth trajectories, appetite regulation, and diet at post-treatment) was explored through group comparisons between the control and treatment groups on weight-for-length scores, subscale scores of the BEBQ, and number of fruits and vegetables consumed in the last week as assessed on a food frequency questionnaire. Prior to between group comparisons, potential differences between the control and treatment group on key sociodemographic and baseline variables (e.g., gender, baseline weight-for-length, household income, caregiver education level) were explored to confirm the effectiveness of randomization to treatment condition. A series of Analysis of Variance (ANOVA) were computed to examine whether the control and treatment groups differed on outcome variables.

Secondary Aim (Determine the feasibility of the HSF intervention and family satisfaction with the treatment) was explored using descriptive analyses. We calculated the average number of treatment sessions attended and the percentage of participants that attended 2 (67%) and 3 (100%) of the sessions. Additionally, we calculated the percentage of caregivers who either "somewhat agree" or "strongly agree" that the intervention was appropriate, timely, helpful, and satisfactory as assessed by the Treatment Satisfaction Survey. Qualitative comments on the Treatment Satisfaction Survey were also reviewed to identify themes regarding additional information to include in the intervention, what information was most helpful, what caregivers would like to see changed about the intervention, and what they would like to see stay the same.